CLINICAL TRIAL: NCT04684186
Title: Real-time Guided Stereotactic Radiotherapy in Lung Cancer Using Endovascular Coils for Tumor Marking: Head-to-head Comparison Between Endovascular and Bronchoscopic Fiducial Marker Insertion
Brief Title: Comparison Between Endovascular and Bronchoscopic Tumor Marker Insertion for Real-time Stereotactic-guided Radiotherapy in Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Rafael DURAN, MD, M.D., Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2016-00046
Record Dates: First submitted 2020-12-07; First posted 2020-12-24 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Lung Cancer; Lung Metastases; Radiotherapy
Keywords: fiducial marker placement; stereotactic body radiotherapy; interventional radiology
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Endovascular fiducial marker insertion: Fiducial markers are inserted and released near the tumor through femoral puncture. A catheter is led through the venous system to the right heart and from there through the heart into the pulmonary arteries.
  Interventions: Procedure: Endovascular fiducial marker insertion
- Bronchoscopic fiducial marker insertion: Fiducial markers are inserted and released near the tumor into the bronchi using an endoscopic route
  Interventions: Procedure: Bronchoscopic fiducial marker insertion

INTERVENTIONS:
Procedure: Endovascular fiducial marker insertion — Fiducial markers will be inserted using an endovascular route
  Groups: Endovascular fiducial marker insertion
Procedure: Bronchoscopic fiducial marker insertion — Fiducial markers will be inserted using an endoscopic route
  Groups: Bronchoscopic fiducial marker insertion

SUMMARY:
The role of radiotherapy is well established in the management of early stage lung cancer or as part of a multidisciplinary approach of locally advanced lung cancer (1).

Recent advances in Cyberknife© technology, which is a robotic system of stereotactic irradiation including localisation and real time lesion-tracking, has led to an increase in accuracy and potentially in efficiency of the irradiation of tumor field (2)(3). According to several studies, promising results in local control and survival rates have been achieved in patients suffering from primary lung cancer or peripheral lung metastasis treated with Cyberknife© (4)(5)(6)(7)(8).

Fiducial markers are implanted in or near a tumor in a configuration defining a COM (center of mass) guiding the Cyberknife for tumor localization.

Tumor movement is then synchronized to respiratory cycle motion during treatment which reduces toxicity of non target lung tissue irradiation. Change in marker positioning leads to COM alterations, thus limiting detection by the tracking system.

Percutaneous (9)(10)(11) (12), endovascular (12)(13) fiducial implantation or by means of bronchoscopic devices (14)(15)(16)(17)(18) are three techniques that have been validated in previous studies as feasible and safe procedures, providing accurate tracking.

Few studies are currently available in the litterature comparing these modalities (19)(20). The percutaneous implantation technique will not be considered for this study because this technique is associated with a high risk of pneumothorax (9).

Both the endobronchial and endovascular technique have been described in the literature with equivalent success rate (87-90%) in intention to treat (21)(22).

One of the endpoints of this study is to verify that these results are reproducible in our institution where both techniques are currently available and to investigate other secondary endpoints such as fiducial marker migration after placement, complications rates and procedure time.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer (primary or secondary, any histological type)
* Early stage lung cancer: patients diagnosed with stage I for which operation is contra-indicated, for example because of cardiac or pulmonary comorbidities.
* Locally advanced lung cancer stages II - IIIB
* Metastatic lung cancer stage IV (palliative care)
* 18 y ≤ age ≤ 85 y

Exclusion Criteria:

* age <18y
* incapacity of judgment
* Absence of a signed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer (1ary and 2ndary), not eligible for surgery, and treated by radiation therapy needing a fiducial marker placement will be eligible for this study which is a prospective randomized controlled trial (endovascular vs endobronchic fiducial marker).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-10-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Cyberknife© tracking | Before Cyberknife
  Tumor tracking assessment by Cyberknife© after bronchoscopic and endovascular fiducial marker implantation

SECONDARY OUTCOMES:
Fiducial implantation evaluation by operator | Immediately post-implantation
  Assessment of technical feasibility of implantation of at least three fiducial markers around the lung tumor in both techniques
Fiducial marker migration | Immediately post-implantation and before Cyberknife
  Secondary fiducial migration rate assessment in both techniques
Procedure time | Immediately after the procedure
  Procedure time required for the implantation of three markers around the lung tumor in both techniques
Complication rate | within 30 days of fiducial marker placement
  Complication rate (AE/SEA) within 30 days of fiducial marker placement in both techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire vaudois - Department of Radiology and Interventional Radiology, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Hagmeyer L, Priegnitz C, Kocher M, Schilcher B, Budach W, Treml M, Stieglitz S, Randerath W. Fiducial marker placement via conventional or electromagnetic navigation bronchoscopy (ENB): an interdisciplinary approach to the curative management of lung cancer. Clin Respir J. 2016 May;10(3):291-7. doi: 10.1111/crj.12214. Epub 2014 Nov 3. PMID 25308297
- [Background] Harada T, Shirato H, Ogura S, Oizumi S, Yamazaki K, Shimizu S, Onimaru R, Miyasaka K, Nishimura M, Dosaka-Akita H. Real-time tumor-tracking radiation therapy for lung carcinoma by the aid of insertion of a gold marker using bronchofiberscopy. Cancer. 2002 Oct 15;95(8):1720-7. doi: 10.1002/cncr.10856. PMID 12365020
- [Background] Siegel R, Ward E, Brawley O, Jemal A. Cancer statistics, 2011: the impact of eliminating socioeconomic and racial disparities on premature cancer deaths. CA Cancer J Clin. 2011 Jul-Aug;61(4):212-36. doi: 10.3322/caac.20121. Epub 2011 Jun 17. PMID 21685461
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] Detterbeck FC, Lewis SZ, Diekemper R, Addrizzo-Harris D, Alberts WM. Executive Summary: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):7S-37S. doi: 10.1378/chest.12-2377. No abstract available. PMID 23649434
- [Background] Detterbeck FC. Lobectomy versus limited resection in T1N0 lung cancer. Ann Thorac Surg. 2013 Aug;96(2):742-4. doi: 10.1016/j.athoracsur.2013.03.074. No abstract available. PMID 23910135
- [Background] Stefani A, Nesci J, Casali C, Morandi U. Wedge resection versus lobectomy for T1N0 non-small cell lung cancer. Minerva Chir. 2012 Dec;67(6):489-98. PMID 23334112
- [Background] Ahn SH, Han MS, Yoon JH, Jeon SY, Kim CH, Yoo HJ, Lee JC. Treatment of stage I non-small cell lung cancer with CyberKnife, image-guided robotic stereotactic radiosurgery. Oncol Rep. 2009 Mar;21(3):693-6. PMID 19212628
- [Background] Shen ZT, Wu XH, Li B, Zhu XX. Clinical outcomes of CyberKnife stereotactic body radiotherapy for peripheral stage I non-small cell lung cancer. Med Oncol. 2015 Mar;32(3):55. doi: 10.1007/s12032-015-0506-1. Epub 2015 Feb 1. PMID 25638468
- [Background] van der Voort van Zyp NC, Hoogeman MS, van de Water S, Levendag PC, van der Holt B, Heijmen BJ, Nuyttens JJ. Stability of markers used for real-time tumor tracking after percutaneous intrapulmonary placement. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):e75-81. doi: 10.1016/j.ijrobp.2010.12.026. Epub 2011 Feb 23. PMID 21349655
- [Background] Patel A, Khalsa B, Lord B, Sandrasegaran K, Lall C. Planting the seeds of success: CT-guided gold seed fiducial marker placement to guide robotic radiosurgery. J Med Imaging Radiat Oncol. 2013 Apr;57(2):207-11. doi: 10.1111/j.1754-9485.2012.02445.x. Epub 2012 Sep 21. PMID 23551782
- [Background] Habermehl D, Henkner K, Ecker S, Jakel O, Debus J, Combs SE. Evaluation of different fiducial markers for image-guided radiotherapy and particle therapy. J Radiat Res. 2013 Jul;54 Suppl 1(Suppl 1):i61-8. doi: 10.1093/jrr/rrt071. PMID 23824129
- [Background] Chan MF, Cohen GN, Deasy JO. Qualitative evaluation of fiducial markers for radiotherapy imaging. Technol Cancer Res Treat. 2015 Jun;14(3):298-304. doi: 10.1177/1533034614547447. Epub 2014 Sep 16. PMID 25230715
- [Background] Pepin E, Olsen L, Badiyan S, Murad F, Mullady D, Wang-Gillam A, Linehan D, Parikh P, Olsen J. Comparison of implanted fiducial markers and self-expandable metallic stents for pancreatic image guided radiation therapy localization. Pract Radiat Oncol. 2015 May-Jun;5(3):e193-e199. doi: 10.1016/j.prro.2014.08.019. Epub 2014 Oct 3. PMID 25413391
- [Background] Boschini FJ, Commander CW, Schreiber EC, Yu H, Dixon RG. Comparison of Gold Seeds, Tight Embolization Coils, and Loose Embolization Coils Used as Fiducial Markers for Dynamic Tracking Using CyberKnife. Pract Radiat Oncol. 2013 Apr-Jun;3(2 Suppl 1):S22. doi: 10.1016/j.prro.2013.01.074. Epub 2013 Mar 25. No abstract available. PMID 24674518
- [Background] Nuyttens JJ, Prevost JB, Praag J, Hoogeman M, Van Klaveren RJ, Levendag PC, Pattynama PM. Lung tumor tracking during stereotactic radiotherapy treatment with the CyberKnife: Marker placement and early results. Acta Oncol. 2006;45(7):961-5. doi: 10.1080/02841860600902205. PMID 16982564
- [Background] Shirato H, Harada T, Harabayashi T, Hida K, Endo H, Kitamura K, Onimaru R, Yamazaki K, Kurauchi N, Shimizu T, Shinohara N, Matsushita M, Dosaka-Akita H, Miyasaka K. Feasibility of insertion/implantation of 2.0-mm-diameter gold internal fiducial markers for precise setup and real-time tumor tracking in radiotherapy. Int J Radiat Oncol Biol Phys. 2003 May 1;56(1):240-7. doi: 10.1016/s0360-3016(03)00076-2. PMID 12694845
- [Background] Chen AP, Setser A, Anadkat MJ, Cotliar J, Olsen EA, Garden BC, Lacouture ME. Grading dermatologic adverse events of cancer treatments: the Common Terminology Criteria for Adverse Events Version 4.0. J Am Acad Dermatol. 2012 Nov;67(5):1025-39. doi: 10.1016/j.jaad.2012.02.010. Epub 2012 Apr 11. PMID 22502948
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Prevost JB, Nuyttens JJ, Hoogeman MS, Poll JJ, van Dijk LC, Pattynama PM. Endovascular coils as lung tumour markers in real-time tumour tracking stereotactic radiotherapy: preliminary results. Eur Radiol. 2008 Aug;18(8):1569-76. doi: 10.1007/s00330-008-0933-x. Epub 2008 Apr 4. PMID 18389249
- [Background] Schroeder C, Hejal R, Linden PA. Coil spring fiducial markers placed safely using navigation bronchoscopy in inoperable patients allows accurate delivery of CyberKnife stereotactic radiosurgery. J Thorac Cardiovasc Surg. 2010 Nov;140(5):1137-42. doi: 10.1016/j.jtcvs.2010.07.085. Epub 2010 Sep 20. PMID 20850809
- [Result] Hong JC, Yu Y, Rao AK, Dieterich S, Maxim PG, Le QT, Diehn M, Sze DY, Kothary N, Loo BW Jr. High retention and safety of percutaneously implanted endovascular embolization coils as fiducial markers for image-guided stereotactic ablative radiotherapy of pulmonary tumors. Int J Radiat Oncol Biol Phys. 2011 Sep 1;81(1):85-90. doi: 10.1016/j.ijrobp.2010.04.037. Epub 2010 Aug 1. PMID 20675070